CLINICAL TRIAL: NCT04487379
Title: Evaluation of Crestal Bone Topography of Edentulous Ridges: A Retrospective Study Comparing Ultrasonography to Cone-Beam Computed Tomography (CBCT)
Brief Title: Ultrasound Crestal Bone Topography of Edentulous Ridges
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Clinical Associate Professor, University of Michigan
Other Study IDs: HUM00183733
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group with edentulous ridge: This group had edentulous ridge planning to receive a dental implant and had ultrasound and cone-beam computed tomography images of the ridge.

SUMMARY:
A successful implant surgery primarily relies on a prudent evaluation of oral anatomy and meticulous treatment planning. Additionally, of paramount importance that dictates the types of procedures, material selection and ultimately success of implant surgery is the quality and quantity of the edentulous ridge. Ultrasound imaging (US), another cross-sectional imaging modality, has been extensively used in the medical diagnostics field. The ability of ultrasound to image soft tissue-bone interface makes it particularly promising for studying bone ridge width and crestal bone topography. Therefore, this retrospective human study aimed to compare bone width measurements between US and CBCT. This study also investigated the possible correlation between the crestal bone surface quality imaged by US and CBCT.

ELIGIBILITY:
Inclusion Criteria:

* Patient records at the Graduate Periodontal Clinic
* With both US and CBCT scans taking within 3 months between each other from Jan 2016 to Mar 2020
* These images had to include at least one edentulous ridge at the anterior, premolar or molar site.
* Multiple sites in a given patient may be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Records of patients who had at least 1 edentulous ridge with a plan for implant placement, had cone-beam computed tomography as standard procedure and ultrasound imaging for off-label use of evaluating the ridge were included.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of ultrasound for estimating ridge width | up to 3 months after image was taken
  measure the edentulous ridge width at 1, 2 and 3 mm apical to the crest on ultrasound images

SECONDARY OUTCOMES:
Accuracy of ultrasound for assessing ridge surface quality | up to 3 months after image was taken
  Evaluate the crestal bone surface quality with ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Not plan to share IPD.